CLINICAL TRIAL: NCT00421109
Title: Double-blind, Randomised, Placebo-controlled, Phase III Study Comparing the Efficacy and Safety of Bilastine 20 mg Once Daily and Levocetirizine 5 mg for the Treatment of Chronic Idiopathic Urticaria
Brief Title: Efficacy Study for the Symptomatic Treatment of Chronic Idiopathic Urticaria
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Faes Farma, S.A. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: BILA 2006/UCI; 2006-001245-33 (EudraCT Number)
Record Dates: First submitted 2007-01-09; First posted 2007-01-11 (Estimated); Last update posted 2012-04-05 (Estimated); Status verified 2012-04

CONDITIONS: Urticaria
Keywords: Urticaria; Hives; Wheals; Flare; Chronic; Idiopathic; Erythema; Skin diseases, vascular; Hypersensitivity, Immediate; Allergic; Cutaneous
MeSH Terms: conditions — Urticaria; Bronchiolitis Obliterans Syndrome; Erythema; Skin Diseases, Vascular; Hypersensitivity, Immediate | interventions — bilastine; levocetirizine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- 1 (Experimental): Bilastine 20 mg
  Interventions: Drug: Bilastine
- 2 (Active Comparator): Levocetirizine 5 mg
  Interventions: Drug: Levocetirizine
- 3 (Placebo Comparator): Placebo
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Bilastine — Encapsulated 20 mg Tablet. Once daily for 28 days
  Arms: 1
Drug: Levocetirizine — Encapsulated 5 mg tablet. Once daily for 28 days
  Other Names: Xyzall
  Arms: 2
Drug: Placebo — Encapsulated tablet. Once daily for 28 days
  Arms: 3

SUMMARY:
The objective of the study is to evaluate the efficacy and tolerability of Bilastine 20 mg Q.D., compared to Levocetirizine 5 mg Q.D. and placebo for the treatment of Chronic Idiopathic Urticaria.

DETAILED DESCRIPTION:
A total of 540 patients with CIU will be enrolled in this pivotal, randomised, multicentre, international, double-blind, placebo and active-comparator controlled, parallel study . Patients will be selected from both public and private clinical practices. The study population includes males and females between 18 and 70 years of age, suffering from CIU for at least 6 weeks prior to entry in the study with no identifiable cause.

ELIGIBILITY:
Inclusion Criteria:

* 18 to 70 years old.
* Documented history of CIU for at least 6 weeks prior to entry in the study.

Exclusion Criteria:

* Dermatological pathology other than chronic idiopathic urticaria.
* History of autoimmune disorders, Hodgkin's disease, lymphoma, leukemia and generalized cancer.
* Pregnant or breast-feeding women.
* Patients who will be operating heavy machinery or need to drive motor vehicles as an essential part of their profession.
* Patients who have a recent history (within previous 12 months) of drug addiction or alcohol abuse.
* Patients who are currently participating in or have participated in another clinical trial within the last 3 months

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 522 (Actual)
Dates: Start 2006-07; Primary Completion 2007-07 (Actual); Study Completion 2007-07 (Actual)

PRIMARY OUTCOMES:
Change from baseline, in the am/pm Total Symptom Score (TSS3), over the 28 days of the treatment period according to the patient's assessment in the diary card. (Reflective Symptoms) | 28 days

SECONDARY OUTCOMES:
Reflective and Instantaneous symptoms scores. | 28 days
QoL questionnaire. | 28 days
Overall assessment of discomfort caused by CIU. | 28 days
Investigator's overall clinical impression. | End of study
Assessment of the Impact of urticaria on the sleep scale. | 28 days

CONTACTS AND LOCATIONS:
Overall Officials: OLMOS, MD, Principal Investigator — HOSP CLINICO SAN CARLOS, SERVICIO DERMATOLOGIA (Madrid- Spain); DE WEERT, MD, Principal Investigator — UZ GENT/ DE PINTELAAN 185 (Belgium); DUBERTRET, MD, Principal Investigator — HOPITAL ST LOUIS/SCE DERMATOLOGIE/1 AV. CLAUDE VELLEFAUX (Paris- France); SIMON, MD, Principal Investigator — UNIV. KLINIKUM LEIPZIG/KLINIK FÜR DERMATOLOGIE (Germany); KAPINSKA-MROWIECKA, MD, Principal Investigator — SZPITAL SPECJALISTYCZNY IM.S. ZEROMSKIEGO/ODDZIAL DERMATOLOGII/ OS. MLODOSCI 11 (Krakow- Poland); BENEA, MD, Principal Investigator — Spit Clin Dermato-Venero."Prof.Dr./Scarlat Longhin"/Calea Serban Voda216,sector4 (Bucharest- Romania); HERRERO, MD, Principal Investigator — CONSULTORIO DE ALERGIA 1° PISO/HOSPITAL JUAN A. FERNANDEZ/CERVINO 3355 (Buenos Aires- Argentina)
Locations (50):
- Argentina (10):
  - Centre nº 101, Buenos Aires
  - Centre nº 105, Buenos Aires
  - Centre nº 104, Buenos Aires
  - Centre nº 103, Buenos Aires
  - Centre nº 107, Buenos Aires
  - Centre nº 109, Buenos Aires
  - Centre nº 108, Buenos Aires
  - Centre nº 100, Mar Del Plata / Buenos Aires
  - Centre nº 106, Rosario - Santa Fe
  - Centre nº 102, Salta
- Belgium (5):
  - Centre nº 202, Aalst
  - Centre nº 200, Edegem
  - Centre nº 201, Ghent
  - Centre nº 204, Ghent
  - Centre nº 203, Kortrijk
- France (6):
  - Centre nº 302, Lyon
  - Centre nº 305, Marseille
  - Centre nº 307, Nice
  - Centre nº 303, Paris
  - Centre nº 308, Quimper
  - Centre nº 301, Reims
- Germany (6):
  - Centre nº 411, Berlin
  - Centre nº 404, Berlin
  - Centre nº 410, Berlin
  - Centre nº 400, Hamburg
  - Centre nº 407, Hanover
  - Centre nº 406, Leipzig
- Poland (8):
  - Centre nº 505, Iwonicz-Zdrój
  - Centre nº 507, Krakow
  - Centre nº 503, Krakow
  - Centre nº 504, Lodz
  - Centre nº 502, Lublin
  - Centre nº 506, Poznan
  - Centre nº 501, Warsaw
  - Centre nº 500, Wroclaw
- Romania (8):
  - Centre nº 704, Brasov
  - Centre nº 700, Bucharest
  - Centre nº 701, Bucharest
  - Centre nº 702, Bucharest
  - Centre nº 705, Bucharest
  - Centre nº 706, Bucharest
  - Centre nº 707, Bucharest
  - Centre nº 703, Craiova Dolj
- Spain (7):
  - Centre nº 804, Vitoria-Gasteiz, Alava
  - Centre nº 802, Badalona, Barcelona
  - Centre nº 801, Leganés, Madrid
  - Centre nº 803, Bilbao, Vizcaya
  - Centre nº 805, Barcelona
  - Centre nº 800, Madrid
  - Centre nº 806, Valencia

REFERENCES:
- [Background] Church MK. Safety and efficacy of bilastine: a new H(1)-antihistamine for the treatment of allergic rhinoconjunctivitis and urticaria. Expert Opin Drug Saf. 2011 Sep;10(5):779-93. doi: 10.1517/14740338.2011.604029. Epub 2011 Aug 11. PMID 21831011
- [Result] Zuberbier T, Oanta A, Bogacka E, Medina I, Wesel F, Uhl P, Antepara I, Jauregui I, Valiente R; Bilastine International Working Group. Comparison of the efficacy and safety of bilastine 20 mg vs levocetirizine 5 mg for the treatment of chronic idiopathic urticaria: a multi-centre, double-blind, randomized, placebo-controlled study. Allergy. 2010 Apr;65(4):516-28. doi: 10.1111/j.1398-9995.2009.02217.x. Epub 2009 Oct 23. PMID 19860762